CLINICAL TRIAL: NCT03517839
Title: The Effect of Inspiratory Muscle Training on Dyspnea Related Kinesiophobia in Chronic Obstructive Pulmonary Disease
Brief Title: Assessment of Impact of Inspiratory Muscle Training on Movement Fear Due to Dyspnea in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Seda Saka, MSc, PT, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: bvusska01
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-02

CONDITIONS: COPD
Keywords: Dyspnea; Inspiratory Muscle Training; Kinesiophobia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental)
  Interventions: Other: Inspiratory muscle trainig
- Control Group (Sham Comparator)
  Interventions: Other: Inspiratory muscle trainig

INTERVENTIONS:
Other: Inspiratory muscle trainig — Inspiratory muscle training in the training group will be administered at least 5 days a week, 15 minutes twice a day, beginning at 30% of the MIP for 8 weeks. Patients will come to the control once a week, the MIP values will be re-measured and the new training intensity will be determined at 30% of the new value. For the control group, a fixed training session will be given for at least 5 days a week, 15 minutes twice a day, not exceeding 15% of the MIP for 8 weeks.

SUMMARY:
In our study, it was aimed to evaluate the effect of inspiratory muscle training on fear of movement due to dyspnea in COPD patients. Participants will be randomly assigned to two groups. Inspiratory muscle training in the training group will be administered at least 5 days a week, 15 minutes twice a day, beginning at 30% of the MIP for 8 weeks. Patients will come to the control once a week, the MIP values will be re-measured and the new training intensity will be determined at 30% of the new value. For the control group, a fixed training session will be given for at least 5 days a week, 15 minutes twice a day, not exceeding 15% of the MIP for 8 weeks.

DETAILED DESCRIPTION:
Pulmonary diseases are a common cause of mortality and morbidity worldwide. Chronic Obstructive Pulmonary Disease (COPD) causes respiratory muscle weakness, but also causes hypercapnia, dyspnoea, oxygen desaturation, and gait disturbances. In COPD, the main symptom is dyspnea and leads to activity limitation. It has been shown that with exercise, the diaphragm workload increases in COPD patients and requires more MIP than healthy humans. This is associated with dyspnea during exercise and tiredness in the respiratory muscles. Dyspnea is defined as the difficulty in breathing of a person. Painful situations are defined as 'kinesiophobia' as a result of physical injuries and fear of repetition of the problem as a result of injury. Similarly, COPD patients avoid themselves from dyspnea-related activities or compensate by reducing the rate of activity. This reduces the severity of the symptom that precedes the symptom that may occur. As a result, fear of movement occurs due to dyspnea. Decrease in the level of activity; social isolation, fear of dyspnea, depression and anxiety result in a stubborn cycle, reducing the quality of life. In order to increase respiratory muscle strength and endurance, to improve the length tension relationship of respiratory muscles and to increase respiratory capacity, respiratory muscle training is performed by using the training principle of skeletal muscles. In COPD, inspiratory muscle training has been shown in many studies to reduce dyspnoea perception, increase exercise capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* FEV1/FVC<%70
* To be able to read and understand Turkish

Exclusion Criteria:

* Having undergone a COPD exacerbation in the last 6 weeks
* Having comorbidities affecting ambulance
* Having cognitive disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Breathlessness Beliefs Questionnaire-BBQ | 3 Minute (before trainig and after training)
  Breathlessness Beliefs Questionnaire-BBQ Breathlessness Perception Questionnaire; is a measure evaluating kinesophobia and anxiety due to the breathlessness of 17 questions answered by one's own practice. Patients score from 1 to 5 (I strongly agree). High scores indicate high levels of kinesiophobia and anxiety due to breathlessness.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf Univercity, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] De Peuter S, Janssens T, Van Diest I, Stans L, Troosters T, Decramer M, Van den Bergh O, Vlaeyen JW. Dyspnea-related anxiety: The Dutch version of the Breathlessness Beliefs Questionnaire. Chron Respir Dis. 2011;8(1):11-9. doi: 10.1177/1479972310383592. Epub 2010 Dec 20. PMID 21172990
- [Result] Beaumont M, Mialon P, Le Ber C, Le Mevel P, Peran L, Meurisse O, Morelot-Panzini C, Dion A, Couturaud F. Effects of inspiratory muscle training on dyspnoea in severe COPD patients during pulmonary rehabilitation: controlled randomised trial. Eur Respir J. 2018 Jan 25;51(1):1701107. doi: 10.1183/13993003.01107-2017. Print 2018 Jan. PMID 29371379